CLINICAL TRIAL: NCT01725698
Title: The Combined Effect of Mesenchymal Stem Cell, HA-CaSO4,BMP-2, and Implant in Inducing The Healing of Critical-Sized Bone Defect
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ismail Hadisoebroto Dilogo, PhD, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SCNONUNION12
Record Dates: First submitted 2012-11-07; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Union
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Stemcell (Experimental): Mesenchymal stem cell, HA-CaSO4, ¬BMP-2, and Implant
  Interventions: Drug: Mesenchymal stem cell, HA-CaSO4, ¬BMP-2, and Implant

INTERVENTIONS:
Drug: Mesenchymal stem cell, HA-CaSO4, ¬BMP-2, and Implant

SUMMARY:
This research is aimed to evaluate the combination of mesenchymal stem cell, HA-CaSO4, BMP-2, and implant in treating critical-sized bone defect.

In the presence of critical-sized bone defect whose defect size is more than 2.5 cm, bone will suffer a healing disturbance. In treating these conditions, the conventional method were vascularised bone grafting and bone transport. But the existing methods of treatment have many weaknesses Vascularized bone graft is a procedure with a high level of difficulty. Hence not every orthopaedic surgeon were able to perform it. It also takes more operating time and its failure rate is also quite high.

Meanwhile, external fixation which is applied with bone transport, was being often complained by the patient in terms of cosmetic and psychologically.

According to diamond concept of bone healing, there are four main factors that influence the bone healing. These factors are osteogenic factor (mesenchymal stem cell), osteconductive factor (HA-CaSO4), osteoinductive factor (bone morphogenetic protein-2) and mechanical component (implant). The potency of each component in fracture healing with/out bone defect has been proved in many studies. The combined effect of these components is often studied as well, but not in critical-sized bone defect.

ELIGIBILITY:
Inclusion Criteria:

* subjects with critical size defect of bone

Exclusion Criteria:

* subjects with patological fracture caused by primary or secondary bone malignancy, imunological deficit, active hepatitis or those who's under immunosuppresant therapy or other therapeutic modality that can interferes with bone healing.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
RADIOGRAPHIC UNION SCALE (RUST Score) as a measure of bone union | Before surgery, after surgery, week 4 , 8, 12, 16, 20, 24 up to 1.5 years
  plain radiograps will be taken to determine whether the bone has healed.

SECONDARY OUTCOMES:
Visual analog scale as the measure of clinical union | Before surgery, after surgery, week 4 , 8, 12, 16, 20, 24 up to 1.5 years
  We will measure VAS (grade 0-10) to determine the clinical union

CONTACTS AND LOCATIONS:
Locations (1):
- University of Indonesia, National University of Singapore, Jakarta, Singapore, Indonesia, Singapore, Indonesia

REFERENCES:
- [Derived] Dilogo IH, Phedy P, Kholinne E, Djaja YP, Fiolin J, Kusnadi Y, Yulisa ND. Autologous mesenchymal stem cell implantation, hydroxyapatite, bone morphogenetic protein-2, and internal fixation for treating critical-sized defects: a translational study. Int Orthop. 2019 Jun;43(6):1509-1519. doi: 10.1007/s00264-019-04307-z. Epub 2019 Feb 12. PMID 30747273